CLINICAL TRIAL: NCT05306288
Title: CASCADE-LUNG: Cancer Screening Assay Using DELFI; A Clinical Validation Study in Lung
Acronym: DELFI-L201
Status: Active, not recruiting | Type: Observational
Sponsor: Delfi Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DELFI-L201
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Lung Cancer Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and may be used to develop and evaluate performance of biomarker assays to detect cancers or other conditions, laboratory process improvements, and proficiency testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Individuals with elevated-risk lung cancer (screening population)
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects enrolled in DELFI-L201 will have blood specimens collected (~30 mL) at enrollment or up to 30 days after enrollment.

SUMMARY:
CASCADE-LUNG is a multisite, prospective, observational, blood specimen collection study in the elevated-risk lung cancer screening population. The primary objective is to demonstrate the performance characteristics, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the DELFI Lung Cancer Screening Test (DLCST).

DETAILED DESCRIPTION:
DELFI identifies circulating tumor DNA (ctDNA) to detect cancer. Participants will be enrolled into the DELFI-L201 study after informed consent and eligibility is confirmed. The study purpose is to validate the performance of the DELFI-based test for the detection of lung cancer among individuals eligible for routine lung cancer screening. Participants will have blood collected and medical record review at baseline and will have medical record reviews at additional timepoints.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

  1. Ability to understand and provide written informed consent
  2. Age ≥ 50 years
  3. Current or former smoker
  4. ≥ 20 pack-years (pack years = number of packs per day × number of years smoked)
  5. An initial or annual follow-up lung cancer screening chest CT planned/scheduled within 30 days after enrollment (i.e., enrollment chest CT scan)

Exclusion Criteria:

* All subjects

  1. Evidence of any diagnosed cancer (including prior lung cancer) other than non-melanoma skin cancer or carcinoma in situ within 2 years prior to enrollment
  2. Prior systemic therapy, definitive therapy, radiation, or surgical resection for any cancer diagnosis within 2 years prior to enrollment (with the exception of surgery for nonmelanoma skin cancer and biopsies)
  3. Any history of hematologic malignancy or myelodysplasia within 2 years prior to enrollment
  4. Any history of organ tissue transplantation
  5. Any history of blood product transfusion within 120 days prior to enrollment
  6. Current pregnancy
  7. Any condition that in the opinion of the Investigator should preclude the participant's participation in the study
  8. Past or current participation in any clinical study sponsored by DELFI Diagnostics or any history of a LDT (Laboratory Developed Test) for early detection of lung cancer by DELFI Diagnostics

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be men and women, current or former smokers, ≥ 50 years of age who are scheduled for a standard-of-care screening chest CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 11935 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics (sensitivity, specificity, PPV, NPV) of the DLCST. | Approximately 24 months

SECONDARY OUTCOMES:
Performance characteristics (sensitivity, specificity, PPV, NPV) of the DLCST. | Up to approximately 36 months
Adverse events (AEs) associated with the blood specimen collection. | Point in time blood collection (1 day) at enrollment

CONTACTS AND LOCATIONS:
Locations (67):
- United States (66):
  - Cullman Clinical Trials, Cullman, Alabama
  - Science 37 (nationwide digital enrollment), Culver City, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - Hoag Hospital, Newport Beach, California
  - Paradigm Clinical Research Center, Inc., Redding, California
  - San Francisco VA, San Francisco, California
  - Clinical Research of California LLC, Walnut Creek, California
  - SCL Health Research Institute, St. Mary's, Grand Junction, Colorado
  - Paradigm Clinical Research Center, Wheat Ridge, Colorado
  - Stamford Health, Stamford, Connecticut
  - Advanced Research, Boynton Beach, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - SIMEDHealth, LLC, Gainesville, Florida
  - Galenus Group, Lehigh Acres, Florida
  - Renstar Medical Research, Ocala, Florida
  - United Medical Research, Port Orange, Florida
  - American Clinical Trials, LLC., Acworth, Georgia
  - Centricity Research Columbus Piedmont, Columbus, Georgia
  - ClinCept, LLC, Columbus, Georgia
  - Coastal Heritage Clinical Research, Hinesville, Georgia
  - Centricity Research Gwinnett Pulmonology, Lawrenceville, Georgia
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Springfield Clinic, Springfield, Illinois
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Ochsner, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Minneapolis VA, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hannibal Regional Healthcare System, Hannibal, Missouri
  - Washington University, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Internal Medicine Associate, Bridgeton, New Jersey
  - CHRISTUS St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Durham VA, Durham, North Carolina
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Northwest Research Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Clinical Research Associates of Central Pa, LLC, DuBois, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Pittsburgh VA Healthcare System, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Ralph H Johnson VA, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - LLM Research, Myrtle Beach, South Carolina
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Greater Heights Memorial Pulmonary and Sleep, Houston, Texas
  - Houston Pulmonary Sleep and Allergy Associates, Houston, Texas
  - North Houston Cancer Clinics, Huntsville, Texas
  - CHRISTUS Trinity Clinic Pulmonary Medicine, Irving, Texas
  - R&H Clinical Research, Inc., Katy, Texas
  - Lumi Research, Kingwood, Texas
  - Central Virginia VA Health System: Hunter Holmes McGuire, Richmond, Virginia
  - UW Medicine Valley Medical Center, Renton, Washington
- Pan American Center for Oncology Trials, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie the results reported in publications of the study may be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan, and informed consent form may also be shared. Data may be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.